CLINICAL TRIAL: NCT04979663
Title: Safety and Efficacy of GEMOX Combined With Donafenib and Tislelizumab as First-line Treatment in Biliary Tract Cancer
Brief Title: GEMOX Combined With Donafenib and Tislelizumab in Biliary Tract Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-07-2310
Record Dates: First submitted 2021-07-27; First posted 2021-07-28 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Biliary Tract Carcinoma
MeSH Terms: interventions — Oxaliplatin; donafenib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Combination of Gemox, Donafenib and Tislelizumab
  Interventions: Combination Product: Combination of Gemcitabine, Oxaliplatin, Donafenib and Tislelizumab

INTERVENTIONS:
Combination Product: Combination of Gemcitabine, Oxaliplatin, Donafenib and Tislelizumab — Combination of Gemcitabine, Oxaliplatin, Donafenib and Tislelizumab every 3 weeks

SUMMARY:
Study design: Prospective, single-arm, single-center study; Primary endpoint: Safety; Secondary endpoints: Disease control rate, overall response rate, conversion rate, overall survival; Main characteristics of enrolled patients: Patients with initially unresectable biliary tract cancer; Interventions: Combination of Gemcitabine, Oxaliplatin, Donafenib and Tislelizumab; Sample size: 10 patients;

Treatment until:

1. successfully conversed to resectable disease
2. progressed disease
3. intolerable toxicity
4. patient requests withdrawal Research process: In this study, patients who met the inclusion criteria were evaluated at the end of every 2 circles of treatment (6 weeks), up to surgical treatment or disease progression.

Safety evaluation: Evaluate adverse reactions according to CTCAE 4.0; Follow up: 12 months after the last case was enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤80 years;
2. ECOG physical condition score: 0~1;
3. Histologically or cytologically confirmed malignant tumor of epithelial origin in the biliary system;
4. Preoperative imaging assessment of the disease stage was III/IV;
5. The main organs function well, and the examination indicators meet the following requirements:

Routine blood tests: Hemoglobin ≥90 g/L (no blood transfusion within 14 days); Neutrophil count ≥1.5×10^9/L; Platelet count ≥80×10^9/L; Biochemical examination: Total bilirubin ≤2×ULN (upper normal value); ALT or AST ≤ 2.5×ULN; Endogenous creatinine clearance ≥ 50 mL /min (Cockcroft-Gault formula); 6. Sign the informed consent voluntarily; 9. Good compliance, and family members willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients with other uncured malignant tumors;
2. Pregnant or lactating women who are required to withdraw from the clinical trial if they become pregnant during the study period;
3. Previous antitumor therapy for the disease in this study;
4. Participated in clinical trials of other drugs within one month;
5. Patients with a known history of other systemic serious diseases before screening;
6. Long-term unhealed wounds or incomplete healing fractures;
7. Previous organ transplantation history;
8. Abnormal coagulation function;
9. Screening for overactivity/venous thrombosis events in the previous year, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism;
10. Having a history of abuse of psychotropic substances and being unable to quit or having mental disorders;
11. A history of immune deficiency or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
12. Concomitant conditions that, in the investigator's judgment, seriously endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Safety: the incidence of adverse events and serious adverse events | 3 weeks
  Incidence of adverse events and serious adverse events

SECONDARY OUTCOMES:
Disease control rate | 6 weeks
  Disease control rate
Overall response rate | 6 weeks
  Overall response rate
Conversion rate | 6 weeks
  Conversion rate
Overall survival | 6 weeks
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Lu Wang, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China